CLINICAL TRIAL: NCT02359838
Title: Patient-Centered Care for the Older Adult With Hematologic Malignancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Gregory A. Abel, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 14-515
Record Dates: First submitted 2015-02-02; First posted 2015-02-10 (Estimated); Results first posted 2022-07-19 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-03

CONDITIONS: Hematologic Malignancy
Keywords: Hematologic Malignancy; Geriatric Assessment; Geriatric Oncology; Frailty
MeSH Terms: conditions — Hematologic Neoplasms; Frailty | interventions — Restraint, Physical

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care (Other): Frail/pre-frail hematologic oncology patients receive usual care
  Interventions: Other: Baseline Geriatric Screening/Assessment
- Geriatrician Co-Management (Active Comparator): Frail/pre-frail hematologic oncology patients receive co-management by a geriatrician
  Interventions: Other: Baseline Geriatric Screening/Assessment; Other: Geriatrician Co-Management

INTERVENTIONS:
Other: Baseline Geriatric Screening/Assessment — All patients receive baseline geriatric screening/assessment by a research assistant to determine frailty status.
Other: Geriatrician Co-Management — A board-certified geriatrician embedded in the oncology clinic will co-manage patients randomized to this arm.
  Arms: Geriatrician Co-Management

SUMMARY:
This research study is evaluating if co-management by a geriatrician embedded in the oncology clinic can improve outcomes for frail older adults with blood cancers. A rigorous pre-entry frailty assessment by a trained research assistant will be followed by randomization to geriatrician co-management versus usual care for patients found to be frail or pre-frail.

DETAILED DESCRIPTION:
Older adults have unique health concerns, and in particular, older adults with blood cancers may have different disease and other health related issues than younger adults with similar diagnoses. One aspect of aging which can make older adults more vulnerable is frailty. Frailty is a general term that describes a decline in multiple areas of health, including the loss of energy, physical ability, and mental ability. Frailty can make it difficult for patients with cancer to respond to treatment and more likely to have side effects. On the other hand, many older patients are not frail despite advanced age. This study is being done to determine if co-management by a geriatrician of older adults who are found to be frail through a detailed baseline assessment can improve outcomes.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 75 and older who present for an initial consultation at the Dana-Farber/Brigham and Women's Cancer Center for hematologic malignancy (transplantation consultation excluded).
* Assessed to be pre-frail or frail on formal baseline geriatric assessment.

Exclusion Criteria:

* Not willing to participate

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 160 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2020-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory A. Abel, MD, MPH, Principal Investigator — Dana Faber Cancer Institute; Jane A Driver, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

REFERENCES:
- See also: Randomized controlled trial of geriatric consultation versus standard care in older adults with hematologic malignancies — https://doi.org/10.3324/haematol.2021.278802

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Usual Care | Geriatrician Co-Management
Started | 100 | 60
Completed | 100 | 48
Not Completed | 0 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Geriatrician Co-Management | Total
Number analyzed (Participants) | 100 | 60 | 160
Age, Customized [Mean (Standard Deviation); unit: years] | 80.3 (3.9) | 80.5 (4.7) | 80.4 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 20 | 56
  Male | 64 | 40 | 104
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Frailty Status [Count of Participants; unit: Participants]
  Pre-Frail | 75 | 49 | 124
  Frail | 25 | 11 | 36

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall Survival at one year
Time Frame: One year
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Geriatrician Co-Management
Number analyzed (Participants) | 100 | 60
Participants | 79 | 49

ADVERSE EVENTS:
Time Frame: 1 year
Description: Adverse events were not collected.
Arm/Group | Usual Care | Geriatrician Co-Management
All-Cause Mortality (participants affected / at risk) | 21/100 | 11/60
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-26): https://cdn.clinicaltrials.gov/large-docs/38/NCT02359838/Prot_SAP_000.pdf